CLINICAL TRIAL: NCT07073547
Title: A Modular, Phase I, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Cellular Kinetics, Immunogenicity, Pharmacodynamics, and Preliminary Efficacy of AZD0120, a Dual-targeting Autologous Chimeric Antigen Receptor T-cell (CAR-T) Therapy Directed Against BCMA and CD19 in Participants With Multiple Myeloma
Brief Title: A Phase I, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Cellular Kinetics, Immunogenicity, Pharmacodynamics, and Preliminary Efficacy of AZD0120 in Participants With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D831EC00001
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; BCMA; CD19; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: AZD0120 will be administrated in one infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0120 (Experimental): AZD0120 will be administrated in one infusion
  Interventions: Biological: AZD0120

INTERVENTIONS:
Biological: AZD0120 — AZD0120 is a BCMA/CD19 dual CAR T cell product under investigation for early-line treatment in subjects with multiple myeloma

SUMMARY:
This is an interventional, modular, open-label, multicenter study to primarily evaluate the safety and tolerability of AZD0120 in adult participants with multiple myeloma (MM).

DETAILED DESCRIPTION:
This modular study aims to evaluate the safety, tolerability, cellular kinetics, pharmacodynamic effect, immunogenicity, and preliminary efficacy of AZD0120 in subjects with newly diagnosed or early relapsed or primary refractory multiple myeloma. Module 1 consists of early line MM (including newly diagnosed MM and early relapsed or primary refractory MM) with AZD0120 (for newly diagnosed multiple myeloma (NDMM), the intervention is with AZD0120 ± maintenance). Module 2 consists of NDMM with AZD0120 ± maintenance.

ELIGIBILITY:
Inclusion Criteria:

Age:

* Males and females ≥18 years of age at the time of consent

Type of Participant and Disease Characteristics:

* Participant must have documented diagnosis of MM per IMWG diagnostic criteria
* ECOG performance status of 0 or 1.
* Adequate organ and bone marrow function.

For NDMM participants:

* Participants on Module 1: Newly diagnosed multiple myeloma (NDMM) without prior anti- myeloma therapy (no more than 2 cycles of induction therapy before enrollment are acceptable)
* For participants on Module 2: Newly diagnosed MM with a maximum of 6 cycles and minimum of 4 cycles of induction therapy completed prior to screening
* Classified as high-risk MM

For Early Relapsed or Primary Refractory MM (1 or 2 prior lines of therapy) participants:

* Have received and failed 1 or 2 lines of anti-myeloma therapy
* Have received a proteasome inhibitor (PI) and immunomodulatory drug (IMiD) as part of their previous therapy
* Have documented evidence of progressive disease based on investigator's determination of response by the IMWG criteria within 1 year of starting treatment, or on or within 6 months of completing treatment of the subject's last line of anti-myeloma therapy, or have confirmed progressive disease within 6 months prior to screening and who are subsequently determined to be refractory or non-responsive to their most recent anti-myeloma treatment regimen

General Exclusion Criteria:

* Have received prior treatment with CAR T therapy directed at any target
* Known active, or prior history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma
* Active or history of plasma cell leukemia at the time of screening
* Seropositive for human immunodeficiency virus (HIV)
* Active Hepatitis B infection
* Active Hepatitis C infection
* Serious underlying medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 2 years
  Incidence and severity of adverse events (AEs)
Serious Adverse Events (SAEs) | 2 years
  Incidence and severity of serious adverse events (SAEs)
Dose Limiting Toxicities (DLT) | 28 days
  Incidence of dose limiting toxicities events

SECONDARY OUTCOMES:
Pharmacokinetic - AUC0-28d, AUCinf, AUClast | 2 years
  Area under the concentration time-curve of AZD0120 level
Pharmacokinetic - Cmax | 2 years
  Maximum AZD0120 level
Pharmacokinetic - Tmax | 2 years
  Time to reach Maximum AZD0120 level
Pharmacokinetic - Clast | 2 years
  Observed concentration of AZD0120 at last quantifiable concentration
Pharmacokinetic - Tlast | 2 years
  Time to last quantifiable concentration of AZD0120 level
Pharmacokinetic - Quantification of CAR transgene levels | 2 years
  Determination of transgene level
Efficacy - Objective Response Rate (ORR) | 2 years
  Defined as proportion of participants who achieve an overall response of PR or better according to the IMWG 2016 criteria
Efficacy - Complete Response Rate (CRR) | 2 years
  Defined as proportion of participants who achieve a CR response or sCR response according to the IMWG 2016 criteria
Efficacy - Minimal Residual Disease (MRD) | 9 months
  Negative rate at 9 months (± 3 months): defined as the proportion of participants with MRD negative status at 9 months (± 3 months)
Efficacy - Duration of Response (DoR) | 2 years
  Defined as the time from first documented confirmed response until date of documented PD per IMWG 2016 criteria or death due to any cause, whichever occurs first
Efficacy - Time to Response (TTR) | 2 years
  Defined as the time from infusion until the date of first documented objective response, as assessed per IMWG 2016 criteria
Humoral Immunogenicity | 2 years
  Prevalence and incidence ADAs against AZD0120 and the impact on PK, efficacy, and safety, as data allow
Module 2 Adverse Events (AEs) Maintenance | 2 years
  Incidence and severity of AEs for maintenance following AZD0120 infusion in participants with NDMM
Module 2 Serious Adverse Events (SAEs) Maintenance | 2 years
  Incidence and severity of SAEs for maintenance following AZD0120 infusion in participants with NDMM

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Duarte, California
  - Research Site, Denver, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org